CLINICAL TRIAL: NCT04729608
Title: A Phase 3, Randomized, Double-Blind, Placebo/Paclitaxel-Controlled Study of Batiraxcept (AVB-S6-500) in Combination With Paclitaxel in Patients With Platinum-Resistant Recurrent Ovarian Cancer (AXLerate-OC)
Brief Title: Batiraxcept (AVB-S6-500)/Placebo in Combination With Paclitaxel in Patients With Platinum-Resistant Recurrent Ovarian Cancer
Acronym: AXLerate-OC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: There were no significant differences in median PFS between batiraxcept + paclitaxel or paclitaxel alone arms. There was no detriment to overall survival. No new safety signals were identified.
Sponsor: Aravive, Inc. (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVB500-OC-004; GOG-3059 (Other: GOG Foundation); ENGOT OV66 (Other: ENGOT); AXLerate-OC (Other: Aravive)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Platinum-resistant Ovarian Cancer
Keywords: Ovarian cancer; Platinum resistant; Recurrent ovarian cancer; High-grade serous adenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Batiraxcept+PAC (Experimental): Combination of batiraxcept and PAC
  Interventions: Drug: Batiraxcept; Drug: Paclitaxel
- Placebo+PAC (Placebo Comparator): Placebo-controlled arm with PAC
  Interventions: Drug: Paclitaxel; Other: Placebo

INTERVENTIONS:
Drug: Batiraxcept — Batiraxcept is an experimental drug
  Other Names: AVB-S6-500
  Arms: Batiraxcept+PAC
Drug: Paclitaxel — Paclitaxel is the standard of care, background therapy
  Other Names: Taxol
Other: Placebo — Matching placebo
  Arms: Placebo+PAC

SUMMARY:
This is a randomized, double-blind Phase 3 study to compare the efficacy and safety of batiraxcept (AVB-S6-500) in combination with paclitaxel (PAC) versus placebo in combination with PAC in patients with platinum resistant recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and documented recurrent ovarian, fallopian tube, or peritoneal cancer. Only patients with high-grade serous adenocarcinoma histology are eligible.
* Aged 18 years or older
* Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 to 1
* Platinum-resistant disease (defined as progression within ≤6 months from completion of most recent platinum-containing regimen and calculated from the date of the last administered dose of platinum therapy).Subject may have been treated with additional regimen(s) subsequent to determination of platinum resistance.
* Available archived tumor tissue or if archived tissue is not available, a fresh tumor biopsy.
* Received at least 1 but not more than 4 prior therapy regimens.

Note: Maintenance therapy OR hormonal therapies should not be counted as a separate therapy.

Note: Patients who have not received prior bevacizumab must be deemed medically inappropriate OR ineligible to receive bevacizumab, refused to receive bevacizumab, or been unable to receive bevacizumab due to lack of access.

* Measurable disease according to RECIST v1.1 criteria
* Normal gastrointestinal function.
* At least 28 days between termination of prior anticancer or hormonal therapy and first administration of batiraxcept.
* Full recovery from all treatment-related toxicities to Grade 1 or less, except alopecia.

Exclusion Criteria:

* Tumors in the breast or bone
* Untreated central nervous system (CNS) metastases. Subjects requiring corticosteroid therapy for the management of their treated CNS metastases may not be on >10 mg/day prednisone or equivalent or have demonstrated signs or symptoms of neurologic instability for 28 days or less prior to randomization.
* Primary platinum-refractory disease (defined as progression during or within 4 weeks after completion of the first platinum regimen)
* Is being treated with concurrent anticancer therapy or other interventional treatments administered for their underlying ovarian cancer.
* Received prior therapy with PAC in the platinum-resistant recurrent setting
* Evidence of clinically significant third spacing (e.g., pleural effusions, ascites, anasarca, etc.) that requires therapeutic intervention within 28 days prior to first dose of batiraxcept/placebo

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Anti-tumor activity of batiraxcept in combination with PAC measured by progression free survival (PFS) in patients receiving batiraxcept + PAC versus patients receiving Placebo+PAC | 4 months
  PFS is the time interval between randomization and radiologically documented disease progression or death, whichever comes first.

SECONDARY OUTCOMES:
Overall survival | 20 months
  Time following the treatment until death

OTHER OUTCOMES:
Duration of response (DOR) | 9 months
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Objective response rate (ORR) | 3 months
  Proportion of subjects who have a confirmed partial or complete response to therapy relative to baseline as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
Incidence of Treatment Emergent Adverse Events (TEAEs) | 10 months
Quality of Life (QOL) | 10 months
  Subject QOL will be assessed using the Functional Assessment Of Cancer Therapy - Ovarian Cancer (FACT-O) questionnaire, which consists of 4 subscales: physical well-being (7 questions), social/family well-being (7 questions), emotional well-being (6 questions), and functional well-being (7 questions), and 12 additional concerns specific to ovarian cancer. All items are rated on a 5 point scale with 0 "not at all" and 4 "very much". The scoring algorithm allows for eight summary scales: the four core well-being subscales, a subtotal of the 27 core items, a subtotal of the 12 ovarian-specific additional concerns, a grand total of the 39 items, and a trial outcome index (sum of the 17 physical and functional wellbeing items plus the 12 ovarian-specific items).
Clinical benefit rate (CBR) | 4 months
Area under the batiraxcept concentration-time curve. | 10 months
Maximum observed batiraxcept concentration. | 10 months
Minimum observed batiraxcept concentration. | 10 months
Pharmacodynamic marker assessment | 10 months
  Change from the baseline in GAS6 serum levels.
Anti-drug antibody (ADA) titers | 10 months
Cancer antigen 125 (CA-125) levels | 10 months

CONTACTS AND LOCATIONS:
Locations (150):
- United States (84):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Disney Family Cancer Center, Burbank, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - UCLA Women's Health Clinical Research Unit, Los Angeles, California
  - UC Irvine Health-Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - University of California, San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Olive View UCLA Medical Center, Sylmar, California
  - Banner MD Anderson Cancer Center/North Colorado Medical Center, Greeley, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - AdventHealth Gynecologic Oncology, Orlando, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Southeastern Regional Medical Center, LLC, Newnan, Georgia
  - Lewis Cancer & Research Pavilion at St. Joseph's/Candler Health System, Inc., Savannah, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Dr. Sudarshan K. Sharma, Ltd., Hinsdale, Illinois
  - Midwestern Regional Medical Center, LLC, Zion, Illinois
  - Community Health Network, Indianapolis, Indiana
  - St Vincent Hospital and Healthcare Center, Indianapolis, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Women's Cancer Care, Covington, Louisiana
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Maine Medical Partners - Women's Health - Division of Gynecologic Oncology, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Beth Israel Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Cox Health, Springfield, Missouri
  - Washington University School of Medicine - Division of Gynecologic Oncology, St Louis, Missouri
  - Mercy Hospital, David C Pratt Cancer Center, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope, Reno, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Optimum Clinical Research Group, LLC, Albuquerque, New Mexico
  - The Blavatnik Family-Chelsea Medical Center at Mount Sinai, New York, New York
  - North Shore Hematology Oncology Assoc. DBA NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke Cancer Center, Durham, North Carolina
  - First Health of the Carolinas, Pinehurst, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University (OSU) Wexner Medical Center OSU Gynecologic Oncology at Mill Run, Columbus, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Kettering Cancer Center, Kettering, Ohio
  - Stephenson Cancer Center - University of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Abington Memorial Hospital, Hanjani Institute for Gyn Onc, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Gynecology Oncology Clinic, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Clinic Gynecology Oncology, Roanoke, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Pro Healthcare Waukesha Memorial Hospital, Waukesha, Wisconsin
- Belgium (8):
  - ZNA Middelheim, Antwerp
  - AZ St Jan Brugge, Bruges
  - UCL St Luc, Brussels
  - AZ Maria Middelares, Ghent
  - UZ Leuven, Leuven
  - CHA Libramont, Libramont
  - CHC Liege, Liège
  - CHU UCL Namur St. Elisabeth, Namur
- Canada (3):
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Clinical Research Unit, Jewish General Hospital, Montreal, Quebec
- China (14):
  - Peking University Cancer Hospital, Beijing, Haidian District
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang, Hangzhou Province
  - Tianjin Cancer Hospital, Tianjin, Hexi District
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Qilu Hospital Of Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang, Shangcheng District, Hangzhou Province
  - The First Affiliated Hospital of Xi 'an Jiaotong University School of Medicine, Xi’an, Shanxi
  - Nantong Tumor Hospital, Nantong, Tongzhou District, Jiangsu Province
  - The Second Hospital of Shanxi Medical University, Taiyuan, Xinghualing District, Shanxi Province
  - Fudan University Shanghai Cancer Hospital, Shanghai, Xuhui District
  - Hunan Cancer Hospital, Changsha, Yuelu District, Hunan Province
  - Sun Yat-sen Memorial Hospital, Guangzhou, Yuexiu District, Guangdong Province
  - Sun Yat-sen University Cancer Center, Guangzhou, Yuexiu District
- Czechia (4):
  - Fakul Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - FN Ostrava-Poruba, Ostrava
  - UG Prague, Prague
- ICANS, Strasbourg, France
- Georgia (6):
  - LTD High Technology Hospital Medcenter, Batumi
  - LTD Tbilisi Oncology, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Consilium Medulla - Multiprofile Clinic, Tbilisi
  - LTD Caucasus Medical Centre, Tbilisi
  - LTD Innova, Tbilisi
- Italy (9):
  - Policlinico S. Orsola-Malpighi - SSD Oncologia Medica, Bologna
  - Ist. di Candiolo - IRCCS Fondazione del Piemonte per l'Oncologia, Candiolo
  - Ospedale "Vito Fazzi" - ASL Lecce, Lecce
  - SC Oncologia - Ospedale San Luca, Lucca
  - IRCCS Ist. Romagnolo per lo studio dei Tumori "Dino Amadori", Meldola
  - IEO - Istituto Europeo di Oncologia, Milan
  - IRCCS, Napoli
  - Nuovo Ospedale Santo Stefano di Prato, Prato
  - Fondazione Policlinico "Agostino Gemelli" IRCCS, Rome
- Poland (5):
  - UCK Centrum Medycyny, Gdansk
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii, Lodz
  - SPSK Nr 2 PUM Klinika Ginekologii Operacyjnej i Onkologii Klinicznej, Szczecin
  - Maria Sklodowska - Curie Instytute Oncolgy Center, Warsaw
- Spain (11):
  - VHIO, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofia (Provincial), Córdoba
  - Hospital General Universitario de Elche, Elche
  - Institut Catala d'Oncologia, Girona
  - ICO, L'Hospitalet de Llobregat
  - Clinica Universidad de Navarra, Madrid
  - Hospital La Paz, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Clinica Universidad de Navarra, Pamplona
  - IVO (Instituto Valenciano de Oncología), Valencia
- United Kingdom (5):
  - Royal United Hospital Bath NHS Foundation Trust, Bath
  - Clatterbridge Cancer Centre, Liverpool
  - The Royal Marsden NHS Foundation Trust (Sutton), London
  - The Royal Marsden NHS Foundation Trust (Fulham Road), London
  - South West Wales Cancer Institute, Swansea

IPD SHARING:
Plan to Share IPD: No